CLINICAL TRIAL: NCT03855475
Title: Mechanical Integrity of Memory Systems in Mild Cognitive Impairment
Brief Title: Aging Brain Structure and Memory in Response to Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: Christiana Care Health Services (Other); University of Illinois at Urbana-Champaign (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1256861; R01AG058853 (NIH)
Record Dates: First submitted 2019-02-14; First posted 2019-02-26 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Mild Cognitive Impairment
Keywords: Exercise; Memory; Brain
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise (Experimental): Exercise training
  Interventions: Behavioral: Aerobic exercise
- Stretching (Active Comparator): Control
  Interventions: Behavioral: Stretching

INTERVENTIONS:
Behavioral: Aerobic exercise — Participants will complete 12 weeks of supervised aerobic exercise, 3 times per week, on a treadmill or stationary bicycle
  Arms: Aerobic exercise
Behavioral: Stretching — Participants will complete 12 weeks of supervised stretching, 3 times per week
  Arms: Stretching

SUMMARY:
This study will measure brain structure through its mechanical properties, assessed with magnetic resonance elastography, and determine whether it improves with aerobic exercise in older adults with low memory abilities. Additionally, this study will determine if memory abilities improve with exercise and if they are related to brain structure. Overall, this project has the potential to identify how brain health is impacted by exercise in older adults.

DETAILED DESCRIPTION:
Mechanical properties of the human brain, measured with magnetic resonance elastography (MRE), reflect the health of brain tissue. Our previous research has shown that these mechanical properties of the hippocampus are highly sensitive to memory function in young adults. Based on these findings, we believe that these mechanical properties may be strong indicators of memory health in older adults and populations experiencing decline in memory function (i.e. mild cognitive impairment, MCI). Further, our results indicate these properties and associated functions are positively impacted by fitness and exercise training, thus making them potentially ideal markers for brain health in assessing rehabilitation.

The objective of this research is to examine these properties in older adults with and without MCI. We will do the following: (1) determine if there are differences in mechanical properties of memory systems in older adults with and without MCI; (2) establish structure-function relationships between mechanical properties and memory performance in the older adult population; and (3) determine if both mechanical properties and memory performance are impacted by cardiovascular health, both through cross-sectional assessment of aerobic fitness and longitudinal response to exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Cognitive function scores consistent with amnestic mild cognitive impairment based on pre-screening evaluation
* age 60-90 years
* MMSE score >24 at time of initial consent

Exclusion Criteria:

* major psychiatric disorder (e.g. schizophrenia, bipolar disorder, major depression within past two years)
* neurological or autoimmune conditions affecting cognition (e.g. Parkinson's disease, epilepsy, multiple sclerosis, head trauma with loss of consciousness greater than 30 min, large vessel infarct)
* other systemic medical illnesses (e.g. cardiovascular disease, cancer, renal failure, diabetes, chronic obstructive pulmonary disease, liver diseases, hypertension)
* current medication use likely to affect CNS functions (e.g. long active benzodiazepines)
* failed outcome on the baseline graded exercise test
* hypertension (systolic 130+ mmHg OR diastolic 80+ mmHg) from baseline blood pressure measurement
* claustrophobia, metal implants, pacemaker or other factors affecting feasibility and/or safety of MRI scanning
* concussion within last 2 years and more than 3 lifetime concussions
* current smoking (including marijuana) within the past 3 months

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change in brain mechanical properties | Baseline, 12 weeks
  Investigators are assessing change in brain structure through mechanical properties in response to exercise from baseline to the end of the 12 week program. An MRI scan with magnetic resonance elastography (MRE) will be used to measure properties of brain regions important to memory (e.g. hippocampus).

SECONDARY OUTCOMES:
Change in relational memory performance | Baseline, 12 weeks
  Behavioral memory test will be used to assess relational memory through accuracy on a spatial reconstruction task.
Change in cardiorespiratory fitness | Baseline, 12 weeks
  Graded exercise test will measure cardiorespiratory fitness through volume of oxygen uptake (VO2)

OTHER OUTCOMES:
Change in brain morphometry | Baseline, 12 weeks
  MRI will be used to measure brain morphometry, i.e. volume
Change in brain function | Baseline, 12 weeks
  MRI will be used to measure brain function, i.e. functional connectivity
Change in brain white matter integrity | Baseline, 12 weeks
  Diffusion MRI will be used to measure integrity of white matter tracts
Change in cognitive function | Baseline, 12 weeks
  NIH Toolbox will be used to assess cognitive function across several domains

CONTACTS AND LOCATIONS:
Overall Officials: Curtis L Johnson, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No